CLINICAL TRIAL: NCT03302936
Title: A Randomized Control Trial Assessing Pyridium for Post-Sling Urinary Retention
Brief Title: Assessing Pyridium for Post-Sling Urinary Retention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Annacecilia Peacher, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GCO 17-0999
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Urinary Retention
Keywords: Midurethral sling; Pyridium
MeSH Terms: conditions — Urinary Retention | interventions — Phenazopyridine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pyridium arm (Experimental): Phenazopyridine 200mg tablet, once prior to surgery
  Interventions: Drug: Phenazopyridine
- Control arm (No Intervention): No intervention in this group. Routine perioperative care.

INTERVENTIONS:
Drug: Phenazopyridine — to be given preoperatively
  Other Names: Pyridium
  Arms: Pyridium arm

SUMMARY:
There has been preliminary data showing that pyridium can decrease the risk of difficulty urinating after midurethral sling. This study is designed to have two groups of patients. One group will receive pyridium pre-operatively, while the other group will have routine preoperative care. Both groups will have their bladder tested prior to going home. It will be evaluated if there is a difference in the difficulty to urinate post-operatively in both groups.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial. It will have two arms with 48 patients in each arm, a total of 98 patients. Patients will be randomized with a block randomization schedule generated by computerized random numbers using a 1:1 allocation to pyridium and routine perioperative care. The study is powered to see a difference in incidence of urinary retention after midurethral sling using 25% as the historic control for our institution. Statistical sample size was based on a decrease in incidence to 5% in the pyridium arm. This is with 80% power and alpha 0.05. After the patient's surgery, including a midurethral sling, the patient will have an active voiding trial performed as described by Pulvino et al. The patient's bladder will be backfilled with 300cc of sterile saline. If the patient cannot tolerate 300cc, the patient will be filled to maximum capacity. The patient will be allowed 20 minutes to void. The patient must void greater than two thirds the volume that was instilled in the bladder to consider it a passed voiding trial. The timing of the voiding trial will be at the discretion of the surgeon, accounting for factors such as complexity of concomitant surgery, the patient being alert, ambulating, with tolerable pain.

ELIGIBILITY:
Inclusion Criteria:

* Any female patient undergoing a midurethral sling surgery, regardless of concomitant pelvic reconstructive or gynecological surgery

Exclusion Criteria:

* Patients with complications from surgery requiring indwelling catheter, bladder/urethral perforation requiring indwelling catheter
* Acute bleeding requiring indwelling catheter for accurate urine output calculation
* Patients undergoing concomitant surgery other than gynecological, preoperative voiding dysfunction defined as postvoid residual >150cc, or spinal anesthesia
* Women who are pregnant, including women of childbearing age who test positive on preoperative urine pregnancy test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 98 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ascher-Walsh, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Arm Vitamin B-6 as Placebo: Vitamin B-6 50mg given once prior to surgery as placebo. Routine perioperative care.
Period: Overall Study
Arm/Group | Pyridium Arm | Control Arm Vitamin B-6 as Placebo
Started | 49 | 49
Completed | 46 | 45
Not Completed | 3 | 4
Not completed — Protocol Violation | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pyridium Arm | Control Arm | Total
Number analyzed (Participants) | 46 | 45 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 29 | 63
  >=65 years | 12 | 16 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 45 | 91
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 13 | 28
  Not Hispanic or Latino | 31 | 32 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 29 | 24 | 53
  More than one race | 15 | 13 | 28
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 46 | 45 | 91
Menopausal status [Count of Participants; unit: Participants] | 22 | 28 | 50
Tobacco user [Count of Participants; unit: Participants] | 7 | 0 | 7
History of abdominal or pelvic surgery [Count of Participants; unit: Participants] | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Considered to Have Passed Their Voiding Trial
Description: Pyridium affect - A patient's bladder is backfilled with water prior to having foley removed. If they can void 200cc of 300cc instilled in the bladder, they are considered to have past their voiding trial.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- Pyridium Arm: Phenazopyridine 200mg tablet, once prior to surgery
  Phenazopyridine: to be given preoperatively
  Failed void trial, 16 participants or 34.5% in the phenazopyridine arm.
- Control Arm: Vitamin B-6 as placebo. Routine perioperative care.
  Failed void trial, 15 participants or 33.3% in the placebo arm.
Arm/Group | Pyridium Arm | Control Arm
Number analyzed (Participants) | 46 | 45
Participants | 30 | 30

2. Primary Outcome: Incidence of Urinary Retention
Description: Incidence of participants that do not pass their voiding trial and go home with an indwelling foley
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- Urinary Retention in Pyridium: Urinary retention is the same value as failed void trial in both arms
- Urinary Retention in Placebo: Urinary retention is the same value as failed void trial
Arm/Group | Urinary Retention in Pyridium | Urinary Retention in Placebo
Number analyzed (Participants) | 46 | 45
Participants | 16 | 15

3. Secondary Outcome: Pain Scale
Description: Pain scale from 0-10. 0-being no pain, 10-being the most pain
Time Frame: Day 1: 6-8 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Pain Scale in Pyridium Arm: At time of void, pain on a VAS scale from 0-10
- Pain Scale in Placebo Arm: At time of void pain on a VAS scale from 0-10
Arm/Group | Pain Scale in Pyridium Arm | Pain Scale in Placebo Arm
Number analyzed (Participants) | 46 | 45
score on a scale | 3 [1 to 4] | 3 [2 to 4]

ADVERSE EVENTS:
Time Frame: Through day of surgery
Groups:
- Pyridium: Phenazopyridine 200mg tablet, once prior to surgery
- Placebo: Vitamin B-6 50mg given once prior to surgery as placebo.
Arm/Group | Pyridium | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/36/NCT03302936/Prot_SAP_000.pdf